CLINICAL TRIAL: NCT02611271
Title: Elimination of Antibiotics During Combined Continuous Renal Replacement Therapy and Cytosorb Adsorptive Therapy in Patients With Sepsis and Acute Kidney Injury
Brief Title: Elimination of Antibiotics During Renal Replacement Therapy and Cytosorb Adsorptive Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, Prof. D. Kindgen-Milles, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2015-11-Studienanmeldung
Record Dates: First submitted 2015-11-03; First posted 2015-11-20 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Critical Illness; Sepsis; Acute Kidney Injury
MeSH Terms: conditions — Critical Illness; Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Piperacillin/Tazobactam: Critically ill patients teated with piperacillin/tazobactam undergoing renal replacement therapy and cytosorb absorption during sepsis
  Interventions: Other: Monitoring of antibiotic drug removal
- Imipenem/Cilastatin: Critically ill patients teated with imipenem/cilastatin undergoing renal replacement therapy and cytosorb absorption during sepsis
  Interventions: Other: Monitoring of antibiotic drug removal

INTERVENTIONS:
Other: Monitoring of antibiotic drug removal — No study specific intervention will be performed

SUMMARY:
Cytokine adsorption using the cytosorb adsorber is currently investigated to reduce the levels of proinflammatory cytokines in patients with severe sepsis and septic shock. The adsorber is frequently used in series with continuous renal replacement therapy. Up to date, no data on the removal of antibiotic drugs during combined renal replacement therapy and cytokine adsorptive therapy is available. Therefore, we want to investigate

- whether and to what extent antibiotic drugs (piperacillin/tazobactam and imipenem/cilastatin) are removed during combined continuous renal replacement therapy and cytosorb adsorption in patients with severe sepsis and septic shock

DETAILED DESCRIPTION:
Patients in this trial are undergoing renal replacement therapy as part of their routine care. Thus, this is an observational trial.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care patients with severe sepsis or septic shock and acute kidney injury requiring continuous renal replacement therapy and cytokine adsorption
* Age > 18 y

Exclusion Criteria:

* < 18 y
* Pregnancy
* Contraindications against citrate-anticoagulation or continuous renal replacement therapy or cytokine adsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients treated for sepsis on surgical intensive care unit undergoing renal replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Removal of antibiotic drugs during the first 8 hours of combined continuous renal replacement therapy and cytosorb adsorption | 8 hours
  Removal of antibiotic drugs during combined CRRT and adsorption will be evaluated by calculating total filter clearance using the drug concentration pre- and postfilter as well as the dialysate concentration. The adsorptive clearance will be evaluated using the pre- and postadsorber concentration. The outcome measure will be removal of antibiotic drug [mg/8 h dosing interval].

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Kindgen-Milles, Prof., Principal Investigator — Department of Anesthesiology, Duesseldorf University Hospital
Locations (1):
- Interdisziplinäre Intensivstation ZOM 1, UKD, Düsseldorf, Germany